CLINICAL TRIAL: NCT07080112
Title: The Impact of Climate Change on Women's Health: A Sustainable Development Goals-Based Peer Education Module
Brief Title: Women's Health & Climate Change: An SDG-Based Peer Education Module
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Beyzanur İşbay Aydemir, Lecturer, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2025/3
Record Dates: First submitted 2025-07-14; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-04

CONDITIONS: Women Health; Climate Change; Nursing Education; Sustainable Development
Keywords: Climate Change; Women's Health; Nursing Education; Sustainable Development Goals; Peer Education

STUDY DESIGN:
Intervention Model Description: The study was designed as a randomized controlled trial. The population consisted of third-year nursing students (84 students) enrolled in the spring semester of the 2024-2025 academic year. The entire population was included in the study. For randomization, the class list of 85 students was used based on their order, and randomization was performed via the website https://www.random.org/ to form the experimental and control groups.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer education (Experimental): The training related to the topic was provided to the students by the Gynecology Nursing intern student group (14 students) from the Nursing Department. The Sustainable Development Goals-Based Peer Education Module was divided into two main sections: reproductive health and environmental factors. Under the reproductive health section, topics included the impact of climate change on adolescence, pregnancy, infertility, and menopause; under the environmental factors section, topics covered nutrition and food security, water and hygiene issues, and the effects of climate change on migrant and refugee women. Data were collected using the Sociodemographic Characteristics Form and the Climate Change Anxiety Scale. Necessary permissions were obtained from the developers of the scales regarding their validity and reliability. The related forms and consent forms were completed by the students before the training, immediately after, and one month after the training.
  Interventions: Behavioral: Peer education
- No intervention (No Intervention): Students in the control group were also provided with the training at the end of the study.

INTERVENTIONS:
Behavioral: Peer education — The study was designed as a randomized controlled trial. The population consisted of third-year nursing students (84 students) enrolled in the spring semester of the 2024-2025 academic year. The entire population was included in the study. For randomization, the class list of 84 students was used based on their order, and randomization was performed via the website https://www.random.org/ to form the experimental and control groups.
  Arms: Peer education

SUMMARY:
In the study, it was aimed to examine the effect of sustainable development goals-based peer education on the effect of climate change on women's health on climate change anxiety levels of students studying in the nursing department of the faculty of health sciences.

DETAILED DESCRIPTION:
Climate change, as a global issue, currently poses numerous negative effects on health. These impacts are particularly profound for certain social groups, such as women. The World Health Organization (WHO) and other health authorities have highlighted the effects of climate change on physical and mental health, nutrition, water security, and public health. Due to biological, social, and economic factors, women are more vulnerable to climate change-related health risks (Dündar & Özsoy, 2020).

Women's specific health periods-such as pregnancy, childbirth, and menopause-can make the challenges posed by climate change even more pronounced. Moreover, climate-related natural disasters, water scarcity, food insecurity, and rising temperatures may hinder women's access to healthcare services and increase health risks for women. This situation necessitates the development of specific strategies and focused attention to improve women's health (İlkin et al., 2020).

In this context, it is crucial for nursing students to develop awareness of the effects of climate change on women's health, as it will play a significant role in their future professional practice. Since nurses are on the front lines of healthcare services, receiving education on this topic will enable them to effectively address public health problems (Küçük Biçer, Acar, & Vaizoğlu, 2015). A peer education program aimed at nursing students seeks to raise awareness of the impact of environmental factors on health and to deepen their understanding of how these factors affect women's health (Parmak & Karaaslan Semiz, 2020; Dündar et al., 2020).

This educational initiative not only teaches nursing students about the health effects of climate change but also contributes to developing strategies to protect women in future healthcare practices. Therefore, this study, titled "The Impact of Climate Change on Women's Health," is considered to hold an important place in nursing education.

Accordingly, this study aims to examine the effect of a peer education intervention on climate change and its impact on women's health on the level of climate change-related anxiety among nursing students studying in the Faculty of Health Sciences.

The study was designed as a randomized controlled trial. The population of the study will consist of third-year nursing students (84 students) enrolled in the spring semester of the 2024-2025 academic year. The entire population will be included in the study. For randomization, the class list of 84 students will be used based on their order, and randomization will be performed using the website https://www.random.org/ to form the experimental and control groups. The relevant trainings will be delivered to the students by the Gynecology Nursing intern student group (14 students) from the Nursing Department.

The Sustainable Development Goals-Based Peer Education Module is divided into two main groups: reproductive health and environmental factors. Under the reproductive health group, topics such as the impact of climate change on adolescence, pregnancy, infertility, and menopause will be covered; under the environmental factors group, topics will include nutrition and food security in climate change, water and hygiene issues related to climate change, and the effects of climate change on migrant and refugee women. Each topic will be planned and presented by two students.

Data will be collected using the Sociodemographic Characteristics Form and the Climate Change Anxiety Scale. Necessary permissions were obtained from the developers of these scales for their validity and reliability. The relevant forms and consent forms will be filled out by the students before the training, immediately after the training, and one month following the training. The control group students will also receive the training at the end of the study.

This research will not be supported by any institution or organization, and the research budget will be covered by the researchers themselves.

Sociodemographic Characteristics Form: Developed by the researchers, this form consists of ten questions including the sociodemographic data of the students.

Climate Change Anxiety Scale (CCAS): Another scale used in this study is the Climate Change Anxiety Scale (CCAS). The scale, consisting of a single dimension with 10 items, was developed by Stewart (2021) and adapted into Turkish by Özbay and Alcı (2021). According to factor analysis results, the Turkish version of the scale has been found to be a valid single-dimension scale. The reliability coefficient (Cronbach's Alpha) was determined as 0.980. The study concluded that the scale is valid and reliable for measuring climate change anxiety among university students in Turkey (Özbay & Alcı, 2021). In this study, the reliability coefficient of the CCAS was found to be 0.934. Additionally, the mean score of the Climate Change Anxiety Scale was determined as 3.1641 out of 5.

Responses to the CCAS were evaluated based on the total scores given for each item. The scale items are rated on a 5-point Likert scale with the options: "Strongly Disagree," "Disagree," "Neutral," "Agree," and "Strongly Agree." The minimum possible score on the scale is 10, and the maximum score is 50. A score closer to 50 indicates a high level of climate change anxiety, whereas a score closer to 10 indicates a low level of anxiety related to climate change.

Inclusion Criteria: All students who were third-year nursing students at the Faculty of Health Sciences and who agreed to participate in the study were included. The reason for including third-year students was that they had taken the Women's Health and Diseases Nursing course in the fall semester and their level of perception on the topic was sufficient.

Assessment Methods Used in the Study: Data were collected using a diagnostic form and the Climate Change Anxiety Scale (CCAS). Participants who decided to join the study were informed in detail about the research by the investigator. Before the interview, the participants were provided with information about the study, and the purpose of the research was explained. After this briefing, written and verbal consent was obtained from the participants confirming their agreement to participate, and the forms were filled out.

Statistical Methods Used in the Study: When evaluating the study data, quantitative variables were presented with descriptive statistics such as mean, standard deviation, median, minimum, and maximum values; qualitative variables were shown using frequency and percentage. For variables showing normal distribution, the Student's t-test was used for comparisons between two groups; One-way ANOVA test was applied for comparisons involving three or more groups, and Bonferroni test was used to identify the group causing the difference. For variables not showing normal distribution, the Mann-Whitney U test was used for comparisons between two groups; the Kruskal-Wallis test was applied for comparisons with three or more groups, and the Dunn test was used to determine the group responsible for the difference. Spearman's correlation analysis was employed to assess relationships between variables. Results were evaluated at a 95% confidence interval with significance at the p<0.05 level.

ELIGIBILITY:
Inclusion Criteria:

* All students who are third-year nursing students in the Faculty of Health Sciences and who consent to participate will be included in the study. The reason for including third-year students is that they have completed the Women's Health and Diseases Nursing course in the fall semester and have an adequate level of understanding of the subject.

Exclusion Criteria:

* Refusing to participate or not providing informed consent Having previously received similar education on climate change or women's health Having a diagnosed serious psychiatric disorder or anxiety disorder that could affect anxiety levels Being unable to attend the training program due to absenteeism or health problems

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-06-05 (Actual); Study Completion 2025-07-14 (Actual)

PRIMARY OUTCOMES:
Climate Change Anxiety Scale (CCAS) | 1 month
  Another scale used in this study is the Climate Change Anxiety Scale (CCAS). This unidimensional scale consists of 10 items and was developed by Stewart (2021) and adapted into Turkish by Özbay and Alcı (2021). According to factor analysis results, the Turkish version of the scale has been confirmed as a valid unidimensional instrument. The reliability coefficient (Cronbach's Alpha) was reported as 0.980. The study concluded that the scale is valid and reliable for measuring climate change anxiety among university students in Turkey (Özbay & Alcı, 2021). In the present study, the reliability coefficient of the CCAS was found to be 0.934. Additionally, the mean score on the Climate Change Anxiety Scale was determined as 3.1641 out of 5.

OTHER OUTCOMES:
Sociodemographic Characteristics Form | 1 month
  Developed by the researchers, this form consists of ten questions containing the students' sociodemographic data.

CONTACTS AND LOCATIONS:
Locations (1):
- Sağlık Bilimleri Ünversitesi, Istanbul, Türkiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://dergipark.org.tr/en/download/article-file/1121538